CLINICAL TRIAL: NCT05175118
Title: Minimally Invasive Surgical Fixation for Unstable Fractures of the Distal End Radius in Adults
Brief Title: Minimally Invasive Fixation for Distal Radius Fractures
Acronym: DRF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdalraouf M Ghozaly, Minimally Invasive Surgical Fixation for Unstable Fractures of the distal end Radius in Adults, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Minimally invasive fixation
Record Dates: First submitted 2021-12-01; First posted 2022-01-03 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimally invasive fixation (Other): Minimally Invasive Surgical Fixation for Unstable Fractures of the distal end Radius in Adults
  Interventions: Device: Minimal invasive surgical fixation of distal radius Fractures

INTERVENTIONS:
Device: Minimal invasive surgical fixation of distal radius Fractures — Fixation of distal radius Fractures by minimal invasive technique

SUMMARY:
Minimally invasive surgery avoids the tissue damage and impairment of physiological function caused by open surgery because of its precise location techniques and can effectively promote the early recovery of wrist function. Under conditions of no cutting of fracture fragments, no blood supply compromise in the fracture fragments

DETAILED DESCRIPTION:
Distal radial fracture is common fracture and internal fixation needed in many cases so we use minimally invasive fixation in this study to minimize open surgery compilations

ELIGIBILITY:
Inclusion Criteria:

1. patients with unstable distal radial fracture
2. skeletally mature Patients.
3. Acute fractures within one weeks of injury

Exclusion Criteria:

1. contaminated open fractures.
2. fractures associated with vascular injury requiring repair, and suspected pathologic Fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Fracture healing | 6 minths
  Rate of fracture healing
Wrist function | One year
  Percentage of restoration of wrist function

SECONDARY OUTCOMES:
Fracture compilations | One year
  Percentage of fracture healing compilations

CONTACTS AND LOCATIONS:
Overall Officials: Ab Ma Ghozaly, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No
Study analytic results

REFERENCES:
- [Background] Liverneaux PA. The minimally invasive approach for distal radius fractures and malunions. J Hand Surg Eur Vol. 2018 Feb;43(2):121-130. doi: 10.1177/1753193417745259. Epub 2017 Dec 12. PMID 29231799
- [Background] Chmielnicki M, Prokop A. [New minimally invasive approach for palmar plating in distal radius fractures]. Z Orthop Unfall. 2015 Feb;153(1):25-8. doi: 10.1055/s-0034-1383103. Epub 2015 Feb 27. German. PMID 25723576
- [Background] Igeta Y, Vernet P, Facca S, Naroura I, Hidalgo Diaz JJ, Diaz JJH, Liverneaux PA. The minimally invasive flexor carpi radialis approach: a new perspective for distal radius fractures. Eur J Orthop Surg Traumatol. 2018 Dec;28(8):1515-1522. doi: 10.1007/s00590-018-2124-z. Epub 2018 Jan 24. PMID 29368237
- [Background] Slutsky DJ. Outcomes assessment in wrist surgery. J Wrist Surg. 2013 Feb;2(1):1-4. doi: 10.1055/s-0033-1333892. No abstract available. PMID 24436782